CLINICAL TRIAL: NCT00112112
Title: A Phase I Randomized, Double-Blind Trial of the Safety and Immunogenicity of FluMist® A Live, Intranasal Influenza Virus Vaccine vs. Placebo in Immunocompromised Children Ages 5 Through 17 Years of Age
Brief Title: Safety Study to Evaluate FluMist in Immunocompromised Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP114
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Cancer
Keywords: cancer, pediatric, influenza, vaccine
MeSH Terms: conditions — Neoplasms; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FluMist (Active Comparator): The total volume of 0.5 mL was administered intranasally with a spray applicator (approximately 0.25 mL into each nostril). Each dose contained approximately 10 to 7th TCID 50 (median tissue culture infectious dose) of each of three influenza virus strains. During the 2005 enrollment period, the three 2004/2005 influenza virus strains were used: A/New Caledonia/20/99(H1N1), A/Wyoming/03/2003(H3N2), and B/Jilin/20/2003). During the 2006 and 2007 enrollment periods, the three 2005/2006 influenza virus strains were used: A/New Caledonia/20/99(H1N1), A/California/7/2004(H3N2), and B/Jiangsu/10/2003 (B/Shanghai/361/2002-like.
  Interventions: Biological: FluMist
- Placebo (Placebo Comparator): Placebo intranasal mist was composed of allantoic fluid stabilized with buffer containing sucrose, potassium phosphate, and monosodium glutamate. The total volume of 0.5 mL was administered intranasally with a spray applicator (approximately 0.25 mL into each nostril).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: FluMist — The total volume of 0.5 mL was administered intranasally with a spray applicator (approximately 0.25 mL into each nostril). Each dose contained approximately 10 to 7th TCID 50 (median tissue culture infectious dose) of each of three influenza virus strains. During the 2005 enrollment period, the three 2004/2005 influenza virus strains were used: A/New Caledonia/20/99(H1N1), A/Wyoming/03/2003(H3N2), and B/Jilin/20/2003). During the 2006 and 2007 enrollment periods, the three 2005/2006 influenza virus strains were used: A/New Caledonia/20/99(H1N1), A/California/7/2004(H3N2), and B/Jiangsu/10/2003 (B/Shanghai/361/2002-like.
  brief description of the arm. This element may not be necessary if the associated intervention descriptions contain sufficient information to describe the arm.
  Arms: FluMist
Biological: Placebo — Placebo intranasal mist was composed of allantoic fluid stabilized with buffer containing sucrose, potassium phosphate, and monosodium glutamate. The total volume of 0.5 mL was administered intranasally with a spray applicator (approximately 0.25 mL into each nostril).
  Arms: Placebo

SUMMARY:
The main purpose of this study is to get information about the safety of a flu vaccine spray, called FluMist, in children with cancer. The study is also being done to find out how much and how long the vaccine spray can be found in the nose.

DETAILED DESCRIPTION:
This study is a randomized, double-blind Phase 1 study of FluMist vs. placebo in mild to moderately immunocompromised children 5 to 17 years of age with cancer. The primary objective of this study is to describe the safety of FluMist compared with placebo in mild to moderately immunocompromised children with cancer. The secondary objectives of this study are to describe the immune responses following vaccination with FluMist and to determine the incidence and duration of viral replication following vaccination with FluMist.

The standard 0.5 mL dose of vaccine or placebo was administered intranasally. Patients were evaluated at four visits scheduled between days 3-5, days 7-10, days 14-28, and days 35-42 for viral shedding via nasal swabs. Safety outcomes were collected at study clinic visits or by telephone contact through 42 days post dose. Serious adverse events and significant new medical conditions were collected through 180 days after receipt of investigational product.

Immune responses were measured by detection of influenza-specific antibodies as measured by the standard hemagglutination inhibition (HAI) assay. Influenza-specific serum antibody isotype levels were determined and nasal swab specimens were analyzed for the expression of influenza-specific immunoglobulin A (IgA). Serum was analyzed for its ability to neutralize viral particles from infecting Madin-Darby canine kidney cells (microneutralization). Baseline immunosuppression as measured by expression of T- and B-lymphocyte subsets was compared to immunosuppression at time points after vaccination. The duration of viral replication and the titers of live-attenuated influenza virus shed was evaluated from nasal swab specimens collected at scheduled time points after administration of FluMist.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 through 17 years of age (not yet reached their 18th birthday) at the time of entry into the study;
* Patient's parent or legal guardian available by telephone during the course of the study;
* Written informed consent (assent if applicable) and Health Insurance Portability and Accountability Act (HIPAA) authorization (if applicable) obtained from the patient's parent or legal guardian;
* Ability of the patient or patient's parent/guardian to comply with the requirements of the protocol;
* Currently receiving chemotherapy and/or radiation therapy for the treatment of cancer or have received chemotherapy in the past 12 weeks;
* If the subject's underlying cancer is a solid tumor, current status must be stable disease, partial response, or complete response to therapy; if the subject's underlying disease is a hematologic malignancy, current status must be in remission;
* Estimated life expectancy of >1 year; and
* Currently has no worse than mild to moderate immunosuppression (meets none of the exclusion criteria).

Exclusion Criteria:

* History of hypersensitivity to any component of FluMist, including egg or egg products, or monosodium glutamate;
* History of hypersensitivity to gentamicin;
* Close contact with a severely immunocompromised patient (e.g., a hematopoietic stem cell transplant patient, during those periods in which the immunocompromised patient requires care in a protective environment);
* History of Guillain-Barré syndrome;
* History of asthma;
* Use of aspirin or salicylate-containing products in the 30 days prior to study vaccination or expected receipt within the study duration;
* Use of anti-influenza medications (including amantadine, rimantadine, oseltamivir, and zanamivir) within 14 days prior to enrollment or expected receipt (unless medically indicated) during this study;
* Currently receiving inhaled steroid therapy;
* Receipt of immunoglobulin within the past 90 days;
* Receipt of stem cell transplant;
* Acute febrile [>100.0°F (37.8°C) oral] illness or acute respiratory illness, e.g., cough or sore throat, within three days prior to enrollment;
* Administration of any live vaccine within 30 days prior to enrollment or if receipt of another live vaccine is expected within 30 days after the vaccination in this study;
* Administration of any inactivated vaccine within two weeks prior to enrollment or if receipt of another inactivated vaccine is expected within two weeks after the vaccination in this study;
* Receipt of an investigational product studied under an investigational new drug (IND) within 10 days prior to study entry or expected receipt of such an investigational product within 10 days after study vaccination (Note: an investigational product not studied under an IND is allowed at the investigator's discretion);
* Pregnancy or, in biologically capable females (e.g., menses within the last year), not willing to agree to acceptable birth control for three months after study vaccination (for those biologically capable, a urine pregnancy test must be performed on the day of vaccination with a negative result);
* Female who is breastfeeding or lactating;
* Any condition or receipt of other medication that, in the opinion of the investigator, might interfere with the evaluation of the vaccine or interpretation of study results;
* At the study screening visit (within 16 days before study vaccination) a CD4+ T cell percentage of <15%;
* At study entry, an absolute neutrophil count less than or equal to 500 cells/mm3;
* Receipt of high-dose systemic corticosteroids (≥ 2 mg/kg total of prednisone or equivalent given daily or on alternating days) for ≥ 14 consecutive days within 30 days prior to or following study vaccination

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raburn Mallory, MD, Study Director — MedImmune LLC
Locations (5):
- United States (5):
  - University of Rochester School of Medicine & Dentistry, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - St. Jude's Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Children's Hospital Regional Medical Center, Seattle, Washington

REFERENCES:
- [Result] Halasa N, Englund JA, Nachman S, Weinberg GA, Huber VC, Allison K, Dubovsky F, Yi T, McCullers JA, Flynn PM. Safety of live attenuated influenza vaccine in mild to moderately immunocompromised children with cancer. Vaccine. 2011 May 31;29(24):4110-5. doi: 10.1016/j.vaccine.2011.03.097. Epub 2011 Apr 13. PMID 21496468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants, 10 in the FluMist group and 10 in the placebo group, were enrolled in the study between 08Aug2005 and 31Mar2008 at 4 sites in the USA.
Pre-assignment Details: A total of 20 participants were randomized in a 1:1 ratio to the FluMist or placebo group. Participants were enrolled on a staggered schedule to assess safety. Four participants were enrolled and treated in 2005, 8 in 2006, and 8 in 2007; each subset was assessed for vaccine-related serious adverse events prior to enrollment of the next subset.
Groups:
- FluMist: The total volume of 0.5 mL was administered intranasally with a spray applicator (approximately 0.25 mL into each nostril). Each dose contained approximately 10^7 TCID 50 (median tissue culture infectious dose) of each of three influenza virus strains.
Period: Overall Study
Arm/Group | Placebo | FluMist
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FluMist | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.2 (3.8) | 12.2 (3.9) | 12.2 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Reactogenicity Events (REs)
Description: Reactogenicity events (REs) are predefined solicited adverse events (AEs) that can potentially occur after vaccine administration. The REs for this study included fever, runny nose/nasal congestion, sore throat, cough, vomiting, headache, muscle aches, chills, tiredness, and irritability.
Time Frame: 0-42 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs. One participant in FluMist group did not have any RE data and was excluded from the RE analysis.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 8 | 9

2. Primary Outcome: Number of Participants Who Had Serious Adverse Events (SAEs)
Description: An SAE is any AE that results in any of the following outcomes: •Death • Life-threatening • Inpatient hospitalization or prolongation of existing hospitalization • Persistent or significant disability or incapacity • Congenital anomaly/birth defect (in the offspring of a study participant) • An important medical event that may may jeopardize the study participant and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 0-180 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: Participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 1 | 3

3. Primary Outcome: Number of Participants Who Had Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigations study participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: 0-42 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
participants | 6 | 10

4. Primary Outcome: Number of Significant New Medical Conditions (SNMCs)
Description: A significant new medical condition is defined as a new diagnosis of a chronic medical condition that does not meet the criteria of a SAE.
Time Frame: 43-180 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: events
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
events | 0 | 0

5. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus
Description: Number of participants with nasal swab samples that contained vaccine-like virus are reported.
Time Frame: 3-5 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
participants | 3 | 0

6. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus
Description: Number of participants with nasal swab samples that contained vaccine-like virus are reported.
Time Frame: 7-10 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
participants | 2 | 0

7. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus
Description: Number of participants with nasal swab samples that contained vaccine-like virus are reported.
Time Frame: 14-28 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

8. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus
Description: Number of participants with nasal swab samples that contained vaccine-like virus are reported. Sample was collected at this time point only if health assessment indicated presence of a respiratory illness, including otitis media.
Time Frame: 35-42 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

9. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus
Description: Number of participants with nasal swab samples that contained vaccine-like virus are reported.
Time Frame: Unscheduled visits occurring during 0-42 days after study vaccination
Population: Participants who received any study vaccine and had any follow-up for REs and/or AEs.
Measure: Number; unit: participants
Units Other Than Participants: participants w/unsched. illness visits
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 0 | 10
Number analyzed (participants w/unsched. illness visits) | 0 | 4
participants |  | 0

10. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Cluster of Differentiation (CD) 19
Description: Mean and standard deviation results of CD19 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: pre-dosing (Day 0)
Population: All randomized participants who received a full dose of study vaccine, had any valid results in the evaluation of immune response, had no protocol deviations, and had the sample available for the specified day were analysed.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
percentage of lymphocytes | 8.6 (7.4) | 4.8 (8.3)

11. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD3
Description: Mean and standard deviation results of CD3 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
percentage of lymphocytes | 83.6 (8.9) | 89.1 (10.3)

12. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD4
Description: Mean and standard deviation results of CD4 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
percentage of lymphocytes | 47.3 (9.8) | 46.7 (7.5)

13. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD8
Description: Mean and standard deviation results of CD8 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
percentage of lymphocytes | 31.4 (8.1) | 38.8 (7.8)

14. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD19
Description: Mean and standard deviation results of CD19 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 8
percentage of lymphocytes | 10.2 (10.8) | 5.1 (8.6)

15. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD3
Description: Mean and standard deviation results of CD3 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 8
percentage of lymphocytes | 82.0 (9.9) | 89.9 (11.6)

16. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD4
Description: Mean and standard deviation results of CD4 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 8
percentage of lymphocytes | 48.2 (11.8) | 46.5 (11.4)

17. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD8
Description: Mean and standard deviation results of CD8 lymphocyte subsets as a percentage of total lymphocytes.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 8
percentage of lymphocytes | 27.9 (8.0) | 39.6 (10.1)

18. Secondary Outcome: Interferon (INF)-Gamma
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 7 | 10
cells per 10^5 T cells | 17.0 (27.2) | 16.5 (25.9)

19. Secondary Outcome: INF-Gamma
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 7 | 10
cells per 10^5 T cells | 28.6 (43.7) | 7.5 (7.6)

20. Secondary Outcome: INF-Gamma
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 7 | 10
cells per 10^5 T cells | 28.0 (38.7) | 16.6 (27.0)

21. Secondary Outcome: Interleukin (IL)-4
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 10
cells per 10^5 T cells | 2.6 (4.3) | 5.5 (8.4)

22. Secondary Outcome: IL-4
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 10
cells per 10^5 T cells | 1.9 (2.7) | 2.6 (3.5)

23. Secondary Outcome: IL-4
Description: Mean and standard deviation spots-forming cells per 10^5 T cells is reported.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^5 T cells
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 10
cells per 10^5 T cells | 2.9 (3.9) | 4.7 (6.1)

24. Secondary Outcome: Human Leukocyte Antigen (HLA) Matched Tetramers CD8+
Description: The antigen-specific response of the T cell populations was measured using HLA-matched tetramers specific for human CD8 cell populations.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 6 | 5
Percentage of lymphocytes | 11.045 (6.452) | 12.778 (6.579)

25. Secondary Outcome: HLA Matched Tetramers CD8+
Description: as for outcome 24
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 6 | 5
Percentage of lymphocytes | 8.048 (6.701) | 8.632 (4.126)

26. Secondary Outcome: HLA Matched Tetramers CD8+
Description: as for outcome 24
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 6 | 5
Percentage of lymphocytes | 7.997 (3.143) | 12.922 (8.607)

27. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Serum Influenza A/H1N1 Hemagglutination Inhibition (HAI) Titers From Baseline to Day 35-42
Description: Participants with a geometric mean fold-rise in influenza-specific nasal HAI titers >= 4 from baseline are reported.
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: All randomized participants who received a full dose of study vaccine, had any valid results in the evaluation of immune response, had no protocol deviations, and had the samples available for the specified days were analysed.
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 1 | 0

28. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Serum Influenza A/H3N2 HAI Titers From Baseline to Day 35-42
Description: Participants with a geometric mean fold-rise in influenza-specific nasal HAI titers >= 4 from baseline are reported.
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 2 | 0

29. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Serum Influenza B HAI Titers From Baseline to Day 35-42
Description: Participants with a geometric mean fold-rise in influenza-specific nasal HAI titers >= 4 from baseline are reported.
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 1 | 0

30. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Influenza A/H1N1 Microneutralization Titers From Baseline to Day 35-42
Description: Participants with a geometric mean fold-rise in influenza-specific nasal microneutralization titers >= 4 from baseline are reported.
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 2 | 0

31. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Influenza A/H3N2 Microneutralization Titers From Baseline to Day 35-42
Description: as for outcome 30
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 2 | 0

32. Secondary Outcome: Number of Participants Who Experienced a >= 4-fold Rise in Influenza B Microneutralization Titers From Baseline to Day 35-42
Description: as for outcome 30
Time Frame: Baseline (pre-dosing on Day 0) and 35-42 days after study vaccination
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
participants | 1 | 0

33. Secondary Outcome: Influenza A/H1N1 Immunoglobulin A (IgA)
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.8 (0.8) | 0.5 (0.0)

34. Secondary Outcome: Influenza A/H1N1 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 3-5 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.8 (0.7) | 0.5 (0.0)

35. Secondary Outcome: Influenza A/H1N1 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1.1 (1.1) | 0.5 (0.0)

36. Secondary Outcome: Influenza A/H1N1 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 14-28 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.9 (0.9) | 1.1 (1.3)

37. Secondary Outcome: Influenza A/H1N1 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1.3 (1.3) | 0.5 (0.0)

38. Secondary Outcome: Influenza A/H3N2 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1.0 (0.8) | 0.7 (0.5)

39. Secondary Outcome: Influenza A/H3N2 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 3-5 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.7 (0.5) | 0.5 (0.0)

40. Secondary Outcome: Influenza A/H3N2 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1.2 (0.8) | 0.7 (0.5)

41. Secondary Outcome: Influenza A/H3N2 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 14-28 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.7 (0.5) | 1.1 (0.9)

42. Secondary Outcome: Influenza A/H3N2 IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1.7 (1.0) | 0.5 (0.0)

43. Secondary Outcome: Influenza B IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.5 (0.0) | 0.5 (0.0)

44. Secondary Outcome: Influenza B IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 3-5 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.5 (0.0) | 0.5 (0.0)

45. Secondary Outcome: Influenza B IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.5 (0.0) | 0.5 (0.0)

46. Secondary Outcome: Influenza B IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 14-28 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.5 (0.0) | 0.5 (0.0)

47. Secondary Outcome: Influenza B IgA
Description: Mean of influenza-specific IgA from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 0.7 (0.5) | 0.5 (0.0)

48. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD56
Description: Mean and standard deviation results of CD56 lymphocyte subsets is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
percent of lymphocytes | 7.6 (5.5) | 5.2 (3.2)

49. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - CD56
Description: Mean and standard deviation results of CD56 lymphocyte subsets is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 8
percent of lymphocytes | 6.6 (5.6) | 4.6 (3.4)

50. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - White Blood Cells
Description: Mean and standard deviation results of white blood cells subsets is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^3/UL
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
cells per 10^3/UL | 3.91 (1.56) | 4.19 (1.49)

51. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - White Blood Cells
Description: Mean and standard deviation results of white blood cells subsets is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cells per 10^3/UL
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 9
cells per 10^3/UL | 4.05 (1.33) | 3.24 (1.10)

52. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Lymphocytes
Description: Mean and standard deviation results of lymphocytes subsets is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
Percentage of lymphocytes | 27.56 (9.25) | 17.62 (7.56)

53. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Lymphocytes
Description: Mean and standard deviation results of lymphocytes subsets is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 9
Percentage of lymphocytes | 23.13 (8.23) | 22.58 (11.89)

54. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Absolute Lymphocytes
Description: Mean and standard deviation results of absolute lymphocytes subsets is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Cells per 10^3/UL
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
Cells per 10^3/UL | 1.03 (0.50) | 0.77 (0.51)

55. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Absolute Lymphocytes
Description: Mean and standard deviation results of absolute lymphocytes subsets is reported.
Time Frame: 7-10 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Cells per 10^3/UL
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 8 | 9
Cells per 10^3/UL | 0.98 (0.57) | 0.77 (0.58)

56. Secondary Outcome: T- and B-lymphocyte Subsets by Flow Cytometry - Absolute Neutrophils
Description: Mean and standard deviation results of absolute neutrophils subsets is reported.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Cells per 10^3/UL
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 7 | 5
Cells per 10^3/UL | 2728.6 (1162.9) | 3300.0 (1534.6)

57. Secondary Outcome: Influenza A/H1N1 Immunoglobulin G (IgG)
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 672.4 (492.8) | 954.7 (1245.3)

58. Secondary Outcome: Influenza A/H1N1 IgG
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 844.0 (645.7) | 924.3 (1207.2)

59. Secondary Outcome: Influenza A/H3N2 IgG
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1842.4 (1989.1) | 799.1 (426.2)

60. Secondary Outcome: Influenza A/H3N2 IgG
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1671.9 (1646.6) | 742.9 (432.2)

61. Secondary Outcome: Influenza B IgG
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 638.6 (334.5) | 599.1 (344.2)

62. Secondary Outcome: Influenza B IgG
Description: Mean of influenza-specific IgG from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 1020.3 (715.6) | 620.2 (472.8)

63. Secondary Outcome: Influenza A/H1N1 Immunoglobulin M (IgM)
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 160.4 (105.4) | 150.1 (107.0)

64. Secondary Outcome: Influenza A/H1N1 IgM
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 134.8 (100.7) | 171.3 (106.7)

65. Secondary Outcome: Influenza A/H3N2 IgM
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 134.7 (100.4) | 153.1 (109.4)

66. Secondary Outcome: Influenza A/H3N2 IgM
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 136.9 (103.1) | 189.9 (98.5)

67. Secondary Outcome: Influenza B IgM
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: pre-dosing (Day 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 72.2 (66.7) | 69.3 (61.0)

68. Secondary Outcome: Influenza B IgM
Description: Mean of influenza-specific IgM from nasal swab is reported. Titers of < 1 were assigned the value of 0.5.
Time Frame: 35-42 days after study vaccination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | FluMist | Placebo
Number analyzed (Participants) | 9 | 10
titer | 68.4 (55.3) | 82.0 (69.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of investigational product administration through Day 42. Serious adverse events were collected from the time of study drug administration through Day 180.
Arm/Group | Placebo | FluMist
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/10
Other Adverse Events (participants affected / at risk) | 9/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | FluMist (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | FluMist (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oral intake reduced (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.The principal investigators (PIs) also agree for data to be presented first as a joint, multi-center publication.